CLINICAL TRIAL: NCT01761188
Title: The Study of CPVI Plus Electrophysiological Substrate Ablation in the Left Atrium During Sinus Rhythm (STABLE-SR) for the Treatment of Persistent Atrial Fibrillation
Brief Title: the Study of STABLE_SR for Persistent Atrial Fibrillation
Acronym: STABLE-SR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Gang Yang, Doctor of Cardiology Department, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201201
Record Dates: First submitted 2012-12-15; First posted 2013-01-04 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Atrial Fibrillation
Keywords: Persistent Atrial fibrillation;LA substrate;ablation;voltage mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STABLE-SR (Experimental): CPVI plus electrophysiologic substrate ablation in the left atrium during sinus rhythm ( STABLE-SR)
  Interventions: Procedure: Ablation
- Control Group (Experimental): conventional stepwise ablation approach for persistent AF(CPVI + Lines +CFE) .
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — electrophysiology substrate mapping is the critical difference between both groups

SUMMARY:
* Background:the ablation outcomes for the treatment of persistent atrial fibrillation are not as satisfactory as paroxsymal AF. The successful rate ranges from 30%-55%. We found a new novel strategy for the modification of LA substrate during sinus rhythm based on our pilot study.
* Hypothesis: our new method may be more effective than conventional strategy.
* Objectives:The primary objective of this investigation is to compare the efficacy of two different AF ablation strategies in patients with persistent AF:Study Group: CPVI plus electrophysiologic substrate ablation in the left atrium during sinus rhythm ( STABLE-SR);Control Group: conventional stepwise approach for persistent AF(CPVI + Lines +CFE) .The secondary objectives of this investigation are to evaluate and compare the safety and procedural characteristics of both groups.
* Sample size: 220
* Time line: 2013 Q1-2014 Q2

DETAILED DESCRIPTION:
what's is STABLE-SR approach? In our center, the LA substrate mapping was performed in patients with paroxysmal AF and persistent AF during sinus rhythm, particularly 20 normal subjects as control group as well. Our study showed that along with the duration of AF the average voltage of LA deceased and the area of low voltage zone increased. The whole activation time of entire LA would be longer. More complex fractionated electrograms was found in LA. Importantly, we identified the low voltage zone (voltage range: 0.1-0.4mV) and the transitional zone (voltage range: 0.4-1.3mV) in which most of complex fractionated electrograms located. Based on our findings a new novel ablation strategy has emerged, which is modification of LA substrate during sinus rhythm (CPVI+STABLE-SR). Our sequential protocol included 5 steps. First CPVI should be completed followed by CTI ablation to be blocked. Then if AF rhythm maintained cardioversion would be taken. High density mapping of LA substrate would be done during sinus rhythm to identify the low voltage zone and transitional zone. Linear ablation or/and spot ablation should be designed according to the mapping results. Finally bidirectional conduction block should be demonstrated for all the linear lesion and all pulmonary veins would be checked for isolation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a first-time ablation procedure for AF;
* Patients with persistent or long-lasting AF; Persistent AF will be defined as a sustained episode lasting > 7 days and less than 1 years; Long-lasting persistent AF will be more than 1 year and less than 5 years.
* Patients must be willing and able to comply with all peri-ablation and follow-up requirements.
* Patients with atrial fibrillation will to accept the procedure of ablation.
* Patients signed the written informed consent for the study.
* Patients can endure the required follow up.

Exclusion Criteria:

* Patients with paroxysmal AF; Paroxysmal AF will be defined as a sustained episode lasting < 7days.
* Patients with contraindications to systemic anticoagulation with heparin or coumadin or a direct thrombin inhibitor.
* Patients with thromboemboli in LAA.
* Patients with left atrial size ≥ 55 mm (2D echocardiography, parasternal long-axis view).
* Patients allergic for contrast or iodine.
* Patients with the SCr >3.5mg/dl or Ccr < 30 ml/min
* Patients with life expectancy < 12 months
* Patients who are in the period of pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-07 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from AF and/or atrial tachyarrhythmias (ATs) off antiarrhythmic drugs (AADs). | 1 year after a single-ablation procedure
  AF and/or AT occurring in the first 3 months after the ablation (blanking period) were censored.Beyond this, any symptomatic or asymptomatic AF or AT episode that lasted for more than 30 seconds was categorized as a recurrence.

SECONDARY OUTCOMES:
total procedure time | 1 year
  time from puncture to the end
fluoroscopy time | 1 year
  total fluoroscopy time
complications | 1 year
  occurrence of serious adverse events that included death, pericardial effusion causing tamponade or requiring pericardiocentesis, cerebrovascular events, significant PV stenosis (symptomatic or asymptomatic ≤70% reduction in PV diameter in ≥1 veins), left atrial-esophageal fistula, diaphragmatic paralysis, and any vascular complication requiring transfusion or intervention

CONTACTS AND LOCATIONS:
Overall Officials: Minglong Chen, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Yu Y, Wang X, Li X, Zhou X, Liao S, Yang W, Yu J, Zhang F, Ju W, Chen H, Yang G, Li M, Gu K, Tang L, Xu Y, Chan JY, Kojodjojo P, Cao K, Fan J, Yang B, Chen M. Higher Incidence of Asymptomatic Cerebral Emboli After Atrial Fibrillation Ablation Found With High-Resolution Diffusion-Weighted Magnetic Resonance Imaging. Circ Arrhythm Electrophysiol. 2020 Jan;13(1):e007548. doi: 10.1161/CIRCEP.119.007548. Epub 2020 Jan 14. PMID 31937118
- [Derived] Yang B, Jiang C, Lin Y, Yang G, Chu H, Cai H, Lu F, Zhan X, Xu J, Wang X, Ching CK, Singh B, Kim YH, Chen M; STABLE-SR Investigators*. STABLE-SR (Electrophysiological Substrate Ablation in the Left Atrium During Sinus Rhythm) for the Treatment of Nonparoxysmal Atrial Fibrillation: A Prospective, Multicenter Randomized Clinical Trial. Circ Arrhythm Electrophysiol. 2017 Nov;10(11):e005405. doi: 10.1161/CIRCEP.117.005405. PMID 29141843